CLINICAL TRIAL: NCT06896968
Title: "Effect of Earthquake Preparedness and Awareness Training on the Preparedness, Earthquake Literacy, and Attitudes Toward Earthquakes of Nursing Students Studying in the First Earthquake Zone
Brief Title: Earthquake Preparedness Training and Nursing Students' Awareness, Literacy, and Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Sabahat Coşkun, Associate Professor Dr., Bilecik Seyh Edebali Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Bilecik18
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Nursing Education; Earthquake Literacy
Keywords: Earthquake Preparedness; Nursing Students; Earthquake Awareness; Earthquake Literacy; Attitudes Toward Earthquakes; Disaster Risk Management

STUDY DESIGN:
Intervention Model Description: The study population consists of nursing students at a university, with the target group being final-year students (n: 105). Final-year students were chosen because they possess a higher level of knowledge and awareness, which enhances their ability to absorb earthquake preparedness and awareness training. Additionally, as future healthcare professionals, they can share this knowledge with others. A power analysis was conducted, assuming a medium effect size (d=0.50) for the intervention's impact on earthquake awareness, preparedness, and attitudes. With α=0.05 and Power=95%, the minimum required sample size was calculated as 54, but the target is to reach 105 students to account for potential dropouts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Earthquake Preparedness and Awareness Training
  Interventions: Behavioral: Earthquake Preparedness and Awareness Training

INTERVENTIONS:
Behavioral: Earthquake Preparedness and Awareness Training — Earthquake Preparedness and Awareness Training + standard education

SUMMARY:
Earthquakes are natural disasters with sudden and destructive effects, causing loss of life, injuries, psychological trauma, and economic losses. Turkey is located on active fault lines, and a significant portion of its population is at risk of earthquakes. Therefore, earthquake preparedness is critically important for public health.

Nursing students, as future healthcare professionals, must be prepared for disasters. Earthquake preparedness and awareness training enable students to act consciously before, during, and after an earthquake, contributing to their effective participation in disaster management. These training programs enhance earthquake literacy, supporting quick and accurate decision-making in high-risk situations.

This study is designed as a non-randomized, pre-test-post-test quasi-experimental study. Data will be collected using the Socio-Demographic Characteristics Form, "Individuals' Knowledge Scale on Readiness Levels Before and During Earthquakes, Individuals' Behavior Scale on Readiness Levels Before and During Earthquakes, Earthquake Literacy Scale, and Attitudes Toward Earthquake Scale." Assessments will be conducted before the intervention and again at the end of a 12-week period following the intervention.

This study aims to comprehensively examine the impact of earthquake preparedness and awareness training on nursing students studying in a high-risk seismic zone in Turkey. Specifically, it will evaluate the students' readiness levels before and during an earthquake, their earthquake literacy, and their attitudes toward earthquakes. By highlighting the significance of educational programs designed to enhance nursing students' knowledge, preparedness, and attitudes toward earthquakes, this research seeks to contribute to strengthening the role of healthcare professionals in disaster management.

DETAILED DESCRIPTION:
Earthquakes are sudden and uncontrollable natural disasters that disrupt societal order, causing loss of life, injuries, severe psychological effects, and economic damage within a short period. Therefore, they are considered a significant public health issue that requires priority attention. Turkey is located on one of the world's most active fault lines, with nearly half of its landmass classified as a first-degree seismic zone. This situation increases the frequency of earthquakes and exposes a large portion of the population to seismic risk.

On February 6, 2023, two major earthquakes struck Turkey, affecting 11 provinces and causing severe loss of life and property. These earthquakes resulted in thousands of fatalities and extensive destruction of homes and businesses. Despite advancements in technology, the precise timing of earthquakes remains unpredictable. However, estimates can be made, and appropriate precautions can significantly reduce the loss of life and property. Preventive measures and conscious interventions taken before an earthquake can help mitigate its devastating effects and protect human life. In this context, the preparedness of healthcare professionals, especially nursing students who represent the future of healthcare, is of utmost importance. As the largest professional group in healthcare, nursing students have the potential to play a crucial role in disaster response.

Being informed and prepared for earthquakes is essential for ensuring the safety of nursing students and protecting public health. Earthquake preparedness and awareness training aim to equip nursing students with the necessary skills to act correctly and effectively before, during, and after an earthquake. Such training enhances earthquake literacy, enabling students to make informed and swift decisions in high-risk situations. Strengthening education on disaster management and emergency healthcare services further supports nurses in taking conscious and effective action during disasters. Research highlights that disaster nursing and management education can reduce mortality, improve healthcare services, and decrease disaster-related costs.

Additionally, earthquake preparedness training positively influences nursing students' attitudes toward earthquakes, encouraging them to take an active role in disaster management. Studies show that individuals with earthquake awareness experience less panic and make more rational decisions during seismic events. Therefore, integrating earthquake preparedness and awareness training into nursing curricula is considered essential. In countries like Turkey, where a significant portion of the population is at risk of earthquakes, it is crucial to enhance the visibility of nurses in disaster response and align their professional roles with contemporary disaster nursing practices. International research indicates that disaster management education increases healthcare professionals' preparedness for emergencies, allowing them to serve their communities more effectively.

This study aims to examine the impact of earthquake preparedness and awareness training on the readiness, earthquake literacy, and attitudes of nursing students studying in a high-risk seismic zone. Implementing an effective training program is expected to enhance students' disaster preparedness levels and play a significant role in protecting public health. The findings of this study are anticipated to contribute to the development of nursing education curricula and the reinforcement of disaster preparedness training.

ELIGIBILITY:
Inclusion Criteria:

* Final-year nursing students
* Students who regularly participate in earthquake preparedness and awareness training
* Students who volunteer to participate in the study

Exclusion Criteria:

* -Students who do not regularly participate in earthquake preparedness and awareness training
* Students who have a diploma or certification in disaster management have not been included.

Exclusion Criteria

* Students who wish to withdraw from the study
* Students who do not attend the training twice during the research process
* Students who do not complete the follow-up period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Earthquake Preparedness Levels Scale for Pre- and During-Earthquake (EPLPDE) | Assessments will be conducted at three time points: at baseline (before training), immediately after training, and at 12 weeks
  This scale was developed in 2023 and has undergone validity and reliability testing. It consists of two separate subscales, which allow for the evaluation of individuals' knowledge and behavior levels regarding preparedness before and during an earthquake. The scale measuring individuals' knowledge level about preparedness before and during an earthquake is answered with "Yes" or "No," with "Yes" receiving 1 point and "No" receiving 0 points. The scale consists of 21 items, with a total score range of 0 to 21, where higher scores indicate a higher level of knowledge regarding earthquake preparedness before and during the event. The scale measuring individuals' behavior level regarding preparedness before and during an earthquake is also answered with "Yes" or "No," where "Yes" receives 1 point and "No" receives 0 points. This subscale includes 18 items, with a score range of 0 to 18, where higher scores indicate a higher level of preparedness behavior before and during the earthquake
Earthquake Attitude Scale | Assessments will be conducted at three time points: at baseline (before training), immediately after training, and at 12 weeks
  This scale was developed in 2023 to assess individuals' attitudes toward earthquakes. It consists of 4 subscales: "Anxiety, Prevention, Neglect, and Fatalism Perception," and includes 41 items. Items 1-11 measure the prevention factor, items 12-32 measure the anxiety factor, items 33-38 measure the neglect factor, and items 39-41 measure the fatalism perception factor. The scale uses a 5-point Likert format (1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree, 5: Strongly Agree). Scores range from 41 to 205. The reliability coefficient of the scale is 0.951.
Earthquake Literacy Scale | Assessments will be conducted at three time points: at baseline (before training), immediately after training, and at 12 weeks
  This scale was developed in 2023. It consists of 3 subscales: Cognitive, Behavioral, and Affective, with 26 items. Items 1-6 measure the cognitive subscale, items 7-17 measure the behavioral subscale, and items 18-26 measure the affective subscale. The scale uses a 5-point Likert format (1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree, 5: Strongly Agree). The lowest possible score is 26, and the highest possible score is 130. A higher score on the scale indicates a higher level of earthquake literacy. The Cronbach's Alpha internal consistency coefficient is 0.896.

CONTACTS AND LOCATIONS:
Overall Officials: SABAHAT COŞKUN, Doç.Dr., Study Director — Bilecik Şeyh Edebali Üniversity
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request, in accordance with ethical guidelines and with participant consent.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Yang F, Wang LH, Zhu RF. Prognostic value of long noncoding RNA TUG1 in human cancers. Minerva Med. 2017 Feb;108(1):101-102. doi: 10.23736/S0026-4806.16.04789-3. No abstract available. PMID 28164690